CLINICAL TRIAL: NCT00751361
Title: Prospective, Randomized, Controlled Clinical Study Evaluating the Efficacy of Rheopheresis for Dry Age-Related Macular Degeneration Dry AMD Treatment With Rheopheresis Trial - ART
Brief Title: Dry Age-Related Macular Degeneration (AMD) Treatment With Rheopheresis Trial
Acronym: ART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Apheresis Research Institute (Other)
Responsible Party: Reinhard Klingel, Prof. Dr., Apheresis Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR-2000
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2008-09

CONDITIONS: Dry Age Related Macular Degeneration
Keywords: Rheopheresis; Dry Age Related Macular Degeneration; AMD; apheresis; microcirculation
MeSH Terms: interventions — Plasmapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Treatment group: Patients receive 10 Rheopheresis treatments within 17 weeks
  Interventions: Device: Rheopheresis / double filtration plasmapheresis
- 2 (No Intervention): No treatment control group

INTERVENTIONS:
Device: Rheopheresis / double filtration plasmapheresis — Rheopheresis is a specific method of therapeutic apheresis, using the methodology of double filtration plasmapheresis.
  Other Names: Rheopheresis; Double filtration plasmapheresis
  Arms: 1

SUMMARY:
Purpose is to evaluate Rheopheresis for the treatment of patients with high-risk dry age-related macular degeneration and no therapeutic alternative. Rheopheresis is a method of therapeutic apheresis using the methodology of double filtration plasmapheresis to treat microcirculatory disorders.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 85 years old
* diagnosis of AMD in both eyes
* must have dry AMD in the study eye
* Study eyes with best-corrected ETDRS-visual acuity of 0.1-0.8
* peripheral veins allowing vascular access to establish the extracorporal circuit.

Exclusion Criteria:

* other retinal or choroidal disorders than AMD
* optic nerve disease, glaucoma
* conditions that limit the view of the fundus
* acute bleeding in any eye

General exclusion criteria for the treatment of Rheopheresis:

* anaemia
* haemorrhagic diathesis or coagulopathy
* diabetes
* serious acute or chronic kidney or liver failure
* hypotension systolic < 100 mmHg
* chronic viral infection (HIV, hepatitis B, C)
* epilepsia, psychosis or dementia
* a malignant disease or any other condition with life expectancy < 12 months
* known history of alcohol or drug abuse and long term serious nicotine abuse

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 1998-11; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome is change in best corrected ETDRS-visual acuity (mean logMar change) after 7.5 months compared to baseline visual acuity for both groups. | 30 weeks (7.5 months)

CONTACTS AND LOCATIONS:
Overall Officials: Frank HJ Koch, Prof. Dr., Principal Investigator — University of Frankfurt
Locations (1):
- University of Frankfurt Department of Ophthalmology, Frankfurt, Germany